CLINICAL TRIAL: NCT06590363
Title: The Effect of Musical Intervention in Anxiety on Patients and Doctors in the Appointment Period
Brief Title: The Effect of Music on Anxiety in the Appointment Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Catia Valesca, Principal Investigator, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 147-2023
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety
Keywords: music; anxiety; heart rate; blood pressure; appointment
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music (Experimental): Corresponded to patients and doctors subjected to the period of listening to zen music in the appointment.
  Interventions: Other: Listening to zen music
- Non-Music (No Intervention): Corresponded to patients and doctors not subjected to the period of listening to zen music.

INTERVENTIONS:
Other: Listening to zen music — We conducted a quasi-randomized controlled clinical trial with two groups: Intervention Group (I), which corresponded to patients and doctors who underwent the period of musical listening in the office; and the Control Group (C), composed of patients and doctors who did not undergo the period of musical listening.
  Arms: Music

SUMMARY:
The goal of this randomized clinical trial is to learn if musical intervention can reduce anxiety on patients and doctors in the appointment period. The main questions it aims to answer are:

Can music reduce the psychological symptoms of anxiety at the end of the appointment? Can music reduce heart rate and blood pressure at the end of the appointment?

Researchers will compare if the presence of zen music during the appointment influences anxiety levels.

Participants in the intervention group will listen to music during the appointment. Those in the control group will not have music in the office during the appointment.

ELIGIBILITY:
Inclusion Criteria:

* scheduled appointment;
* agree to participate in the clinical trial.

Exclusion Criteria:

* 17 years or younger;
* deaf;
* illiterate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Anxiety | 16 weeks
  Participants achieved a response if they scored of the State-Trait Anxiety Inventory reduze in the end of the appointment.
  STAI scores are classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

SECONDARY OUTCOMES:
Heart rate | 16 weeks
  Participants achieved a response if the heart rate reduze in the end of the appointment
Blood Pressure | 16 weeks
  Participants achieved a response if the systolic and diastolic blood pressure reduze in the end of the appointment

CONTACTS AND LOCATIONS:
Locations (1):
- Cátia Valesca Nunes Solis, Coimbra, Coimbra District, Portugal